CLINICAL TRIAL: NCT01829178
Title: Phase 2-3 Study of Silymarin on Cisplatin Induced Nephrotoxicity
Brief Title: Evaluation of Effects of Silymarin on Cisplatin Induced Nephrotoxicity in Upper Gastrointestinal Adenocarcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91-03-33-18878
Record Dates: First submitted 2013-01-11; First posted 2013-04-11 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Upper GI Cancer; Cisplatin Adverse Reaction
Keywords: cisplatin; nephrotoxicity; antioxidant; urine neutrophil gelatinase-associated lipocalin (NGAL)
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Silymarin; milk-thistle extract; Drug Therapy; Cisplatin; Fluorouracil; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Placebo Comparator): Placebo 420 mg daily in three divided doses for 65 days as control along with [cisplatin 50-60mg/m2 + fluorouracil 750 mg/m2 +docetaxel 60-80 mg/m2]
  Interventions: Drug: Placebo; Drug: chemotherapy
- Exprimental: Silymarin and chemotherapy (Active Comparator): silymarin 420 mg daily in three divided doses for 65 days along with standard chemotherapy [cisplatin 50-60mg/m2 + fluorouracil 750 mg/m2 +docetaxel 60-80 mg/m2 control
  Interventions: Drug: Silymarin; Drug: chemotherapy

INTERVENTIONS:
Drug: Silymarin — Silymarin 420 mg in 3 divided dose plus standard chemotherapy
  Other Names: Milk thistle
  Arms: Exprimental: Silymarin and chemotherapy
Drug: Placebo — placebo tablets: 420 mg in 3 divided dose
  Other Names: Identical inert tablet to mimic silymarin (140 mg)
  Arms: Control arm
Drug: chemotherapy — All patients will receive standard chemotherapy: cisplatin 50-60mg/m2 + fluorouracil 750 mg/m2 + docetaxel 60-80 mg/m2
  Other Names: Cisplatin; fluorouracil; Docetaxel

SUMMARY:
Cisplatin is a potent chemotherapeutic agent that has been widely used to treat many solid tumours. acute renal failure, despite conservative fluid and electrolyte management, frequently reported adverse event and limiting cisplatin use. Silymarin, a flavonolignan complex isolated from Silybum marianum, has a strong antioxidant, hepatoprotective, anticancer and in animal model nephroprotective properties. Neutrophil gelatinase-associated lipocalin (NGAL) protein is a promising biomarker to detect acute kidney injury due to cisplatin. Milk thistle extract inhibitory effects on epidermal growth factor receptor, vascular endothelial growth factor and insulin-like growth factor-I have shown in the previous in-vitro studies.The aim of present study,a randomized double-blind placebo- controlled clinical trial, to investigate the therapeutic effect of silymarin on cisplatin induced nephrotoxicity and it's impact on chemotherapy. Fifty-eight patients with diagnosed upper gastrointestinal tract carcinomas randomized to silymarin (420mg) or placebo plus chemotherapy [cisplatin 50-60 mg/m2, 5-fluorouracil mg/m2, docetaxel 60-80 mg/m2 every 21 days] for 63 day after inclusion. serum creatinin, blood urea nitrogen (BUN), serum and urine electrolyte will be measured daily during chemotherapy.

changes in urine NGAL, serum vascular endothelial growth factor (VEGF)and caspase activity assessed up to 64 days.

DETAILED DESCRIPTION:
This study will look for possible protective effects silymarin on kidney injury in patients receiving cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* diagnosed
* measurable upper gastrointestinal adenocarcinoma
* swallow problem
* would like to participate in the study
* Glomerular filtration rate(GFR)>45ml/min/1.73m2

Exclusion Criteria:

* end stage renal disease
* requiring dialysis
* post transplantation
* receiving contrast media during last 72 hours
* chronic use of corticosteroids
* chronic use of angiotensin-converting enzyme inhibitor(ACEI )
* untreated hypo-and hyperthyroidism
* ejection fraction<60%
* active urinary tract infection
* iver disease ( five fold increase of liver enzyme in asymptomatic or 3 fold increase in symptomatic
* use of other nephrotoxic agents such as aminoglycoside, amphotericin
* karnofsky performance status <70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Urine concentration of NGAL | up to 9 weeks
  All subject receive silymarin at dose of 420mg or placebo in three dose for 65 consecutive day, urine NGAL concentration will be measured.

SECONDARY OUTCOMES:
Changes in VEGF Serum concentration | up to 9 weeks
  To assess interaction between silymarin and cancer chemotherapy serum vascular endothelial growth factor will be measured.
Tissue activity of caspase 3 | up to 9 weeks
  To assess interaction between silymarin and cancer chemotherapy Tissue activity of caspase 3will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Simin Dashti-Khavidaki, Dr, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Science, Tehran, Tehran Province, Iran